CLINICAL TRIAL: NCT05313529
Title: Effects of Liraglutide, Empagliflozin and Linagliptin on Mild Cognitive Impairment Remission in Type 2 Diabetes (LIGHT-MCI): A Multicentre, Randomised Controlled Trial With An Extension Phase
Brief Title: LIGHT-MCI Trial: GLP-1 Agonist, SGLT2 Inhibitor, and DPP-4 Inhibitor for MCI Remission in Type 2 Diabetes
Acronym: LIGHT-MCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Nanjing First Hospital, Nanjing Medical University (Other); The Affiliated Jiangning Hospital of Nanjing Medical University (Other); Wuxi People's Hospital (Other); Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-ZD-03
Record Dates: First submitted 2022-03-19; First posted 2022-04-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus; Mild Cognitive Impairment
Keywords: Functional MRI; cognition; Olfactory function; Liraglutide, Empagliflozin and Linagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — Liraglutide; Metformin; empagliflozin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liraglutide (Experimental): Liraglutide will be titrated from 0.6mg/day to a final dose 1.8mg/day during the first 2 weeks, if well tolerated.
  Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 8-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but liraglutide could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Liraglutide
- Empagliflozin (Experimental): Empagliflozin will be initiated and maintained at 10mg/ day every morning until the completion of the study.
  Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 8-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but Empagliflozin could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Empagliflozin
- linagliptin (Experimental): linagliptin will be initiated at 5mg/ day every morning. Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 8-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but linagliptin could not be adjusted.
  If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be titrated from 0.6mg/day to 1.8mg/day during the first 2 weeks, if well tolerated. All patients will also continue on their existing dose and regimen of metformin throughout the study
  Other Names: metformin
  Arms: Liraglutide
Drug: Empagliflozin — Empagliflozin will be initiated and maintained at 10mg/ day every morning until the completion of the study. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Empagliflozin
Drug: Linagliptin — Iinagliptin will be initiated at 5mg/ day every morning until the completion of the study. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: linagliptin

SUMMARY:
This is an investigator-led prospective, randomized, open label, parallel study to explore and evaluate the therapeutic effects of Liraglutide, Empagliflozin and Linagliptin on the cognitive function in T2DM patients with mild cognitive impairment (MCI), consisting of a 48-week core study followed by a 28-week extension phase.

DETAILED DESCRIPTION:
The LIGHT-MCI trial is an investigator-led, prospective, randomized, open label, parallel, multi-center study to explore and evaluate the therapeutic effects of Liraglutide, Empagliflozin and Linagliptin on the MCI remission in T2DM patients with MCI inadequately controlled with metformin monotherapy. The trial consists of a 48-week core study followed by an extension phase through to 76 weeks and the investigators will screen in the outpatient and inpatient departments to enroll 396 patients (132 for each arm) totally with the inclusion and exclusion criteria. The patients will be randomized at a 1:1:1 ratio into Liraglutide, Empagliflozin and Linagliptin treatment group with a computer-generated random order. All patients will also continue on their existing dose and regimen of metformin throughout the study. At the baseline, clinical information collection, 100g-steamed bread meal test, biochemical measurement, body composition analysis, cognitive assessment, olfactory test and functional magnetic resonance imaging(fMRI) scan will be conducted for all patients. During the treatment period, visits at 8-week intervals will be performed to evaluate the safety of drugs and adjust the dose of metformin if hypoglycaemia occurs; meanwhile, fasting and 2-hour postprandial plasma glucose assayed by fingerstick, physical examination, and olfactory test will be conducted. Participants who complete the 48-week core study will have the option to receive an additional 28 weeks of intervention after signing an extension consent form. At 48 and 76 weeks of treatment, all of the assessments will be performed again for all recruited subjects, including early withdrawal patients.

ELIGIBILITY:
Inclusion criteria

1. Participants aged ≥40 and ≤75 years, of any gender.
2. Type 2 diabetes diagnosed according to the American Diabetes Association criteria
3. Mild cognitive impairment diagnosed according to the established criteria

   1. Cognitive concern from the patient, or an informant or skilled clinicians
   2. Objective evidence of cognitive impairment: education-adjusted MoCA score ≤ 25 and ≥ 18; or ≥1.0 standard deviation below the mean of age- and education-specific groups on any cognitive subdomain
   3. Preservation of independence in daily living abilities: Barthel Index score ≥ 60
   4. Absence of dementia
4. Treatment with a stable glucose lowering regimen of metformin monotherapy (≥ 1,000 mg daily) or combination with sulfonylurea/glibenclamide/glycosidase inhibitor/basal insulin over the previous 3 months
5. Glycosylated hemoglobin (HbA1c) during screening between ≥7.0% and ≤10.0%
6. BMI of ≥ 19 kg/m2
7. Education duration of ≥6 years
8. Right-handed participants
9. Understanding of the research procedures and methods, potential benefits and risks of the trial, and sign written informed consent

Exclusion criteria

1. History of other dementia-related neurological diseases, depression within the past 2 years, developmental disorders, mania, depression, schizophrenia, etc.
2. Significant nasal sinusitis, nasal cavity and sinus polyps, cranial or nasopharyngeal tumors and other space-occupying lesions, congenital diseases and trauma of the nose, maxillofacial area, and skull base that affect olfaction. Symptoms of upper respiratory tract infection on the day of MRI examination, including nasal congestion, rhinorrhea, fever, etc.
3. Acute metabolic complications such as diabetic ketoacidosis, hyperglycemic hyperosmolar state and hypoglycemic coma within the previous 6 months
4. Severe organ dysfunction of heart, liver, kidneys, and thyroid, including unstable angina, myocardial infarction, or grade II and above cardiac insufficiency within 3 months before screening; estimated glomerular filtration rate (eGFR) by CKD-EPI formula <45 mL/min/1.73 m², alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater exceeding twice the upper limit of normal, hyperthyroidism or uncontrolled hypothyroidism
5. History of medullary thyroid carcinoma, pancreatitis, multiple endocrine neoplasia syndrome type 2, recurrent urinary tract infections, severe gastrointestinal diseases or history of gastrointestinal surgery, history of malignant tumors
6. With MRI contraindications, such as implanted metal prosthesis, claustrophobia, etc.
7. Females who are pregnant, lactating, breast feeding or of child bearing age without effective contraception
8. Participated in other clinical trials within the previous 6 months
9. Known or suspected allergy to the study drugs
10. Received treatment with GLP-1RAs, dual GLP-1R/GCGR agonist, SGLT-2 inhibitors or DPP4 inhibitors in the past 3 months
11. Known history of drug or alcohol abuse within the past 6 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Mild cognitive impairment (MCI) remission rate | The core study spans from baseline to 48 weeks
  MCI mitigation is defined by three criteria: an education-adjusted score of the Montreal Cognitive Assessment (MoCA) ≥26, no cognitive deficits in any explored cognitive subdomain, including processing speed, executive function, immediate memory, visuospatial construction ability, language, attention and delayed memory, evaluated by Trail-Making Test, Stroop Color-Word Test and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), respectively, and preservation of ability to perform instrumental activity of daily living (IADL) with a Functional Activities Questionnaire (FAQ) score <5.

SECONDARY OUTCOMES:
Change in score of Mini-Mental State Examination (MMSE) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The MMSE contains a total of 30 items that assess orientation, registration, attention and calculation, recall, and language, with a score range from 0 to 30. Generally, a higher MMSE score reflects a better cognitive function.
Changes in score of MoCA | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The MoCA (Chinese version) is a screening instrument for MCI comprised of 30 items to assess multiple cognitive domains (memory recall, visuospatial abilities, executive functions, attention, language, and orientation to time and place; scores range from 0 to 30, with higher scores indicating better cognitive function). Participants received one additional point if they had a MoCA score < 30 and 12 years or less of formal school education.
Changes in total score of RBANS | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The RBANS (Chinese version) is a brief neuropsychological screening battery with established test-retest reliability and age-appropriate normative data, which consists of 12 task tests assessing 5 cognitive domains, namely immediate memory, visuospatial/ constructional, language, attention and delayed memory, with a score range from 40 to 160. A higher RBANS score reflects a better global cognitive function.
Change in the RBANS index score of immediate memory | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The RBANS (Chinese version) is a brief neuropsychological screening battery with established test-retest reliability and age-appropriate normative data. The RBANS includes 12 sub-tests that generate five age-adjusted index scores and a total score. The five indices include immediate memory (consisting of list learning and story memory tests), visuospatial/constructional domain (consisting of figure copying and line orientation tests), language (consisting of picture naming and semantic fluency tests), attention (consisting of digit span and coding tests) and delayed memory (consisting of list recall, story recall, figure recall and list recognition tests). Generally, a higher index score reflects a better cognitive subdomain function.
Change in the RBANS index score of visuospatial/constructional | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as the RBANS index score of immediate memory.
Change in the RBANS index score of language | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as the RBANS index score of immediate memory.
Change in the RBANS index score of attention | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as the RBANS index score of immediate memory.
Change in the RBANS index score of delayed memory | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as the RBANS index score of immediate memory.
Change in aggregate time to test completion for Trail Making Test (TMT) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The TMT is a validated timed measure of processing speed, which consists of part A and part B (TMT-A and TMT-B). The time limits for performing the TMT-A and TMT-B are 180 and 300 seconds, respectively. Processing speed is estimated by the aggregate time in seconds to complete TMT-A and TMT-B such that less time indicate faster processing speed.
Change in aggregate time to test completion for Victoria Stroop Color-Word Test | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The Victoria Stroop Color-Word Test is a well-known measure of executive function. There are three indices including Stroop-dot, Stroop-word and Stroop-color word in the test. The color task consists of colored dots; the word task comprises ordinary words that are unrelated to the meaning of color; the color-word task consists of words written in color that indicate the meaning of the color, but the color of these words differs from the meaning of the word itself. The participants were asked to quickly read the color of the dots or Chinese words on the cards. The sum of consuming time taken to read the three cards is used as an index of executive function performance. Less time indicates better executive function.
Changes in MRI-derived total brain volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Philips TX 3.0T superconducting clinical MRI will be used for magnetic resonance scanning (Philips Achieva 3T TX Medical Systems, Eindhoven, the Netherlands). T1 images were processed using Freesurfer software (version 8.1.0, https://surfer.nmr.mgh.harvard.edu) to calculate intracranial volume, total gray matter volume, total white matter volume, cerebrospinal fluid volume and volumes of 68 cortical and 14 subcortical regions based on the Desikan-Killiany atlas23. The total brain volume was calculated as the sum of the gray matter and white matter volumes.
Changes in MRI-derived total gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived total white matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived cerebrospinal fluid volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived white matter hyperintensity volume (WMH) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Total white matter hyperintensity volume was measured from FLAIR images using the Lesion Segmentation Tool for Statistical Parametric Mapping (SPM) 12.0.
Changes in MRI-derived frontal gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume. Frontal gray matter volume was calculated as the sum of all frontal lobe regions parcellated by FreeSurfer (Desikan-Killiany atlas).
Changes in MRI-derived parietal gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume. Parietal gray matter volume was calculated as the sum of all parietal lobe regions parcellated by FreeSurfer (Desikan-Killiany atlas).
Changes in MRI-derived temporal gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume. Temporal gray matter volume was calculated as the sum of all temporal lobe regions parcellated by FreeSurfer (Desikan-Killiany atlas).
Changes in MRI-derived occipital gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume. Occipital gray matter volume was calculated as the sum of all occipital lobe regions parcellated by FreeSurfer (Desikan-Killiany atlas).
Changes in MRI-derived insula gray matter volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived hippocampal volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived parahippocampal volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived entorhinal cortex volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived inferior parietal lobule volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived precuneus volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived cuneus volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived thalamus volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived caudate nucleus volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived putamen volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived pallidum volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived amygdala volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in MRI-derived accumbens volume | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurements and instruments are the same as total brain volume.
Changes in mean fractional anisotropy (FA) in white matter derived from diffusion tensor imaging (DTI) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Diffusion Toolbox in FMRIB Software Library (FSL, version 6.0.7, http://fsl.fmrib.ox.ac.uk/fsl/fslwiki) was used to process all DTI-scans, and generate FA maps. FA from DTI assessment is a global microstructural integrity measure, with higher value indicating better integrity.
Changes in mean diffusivity (MD) in white matter derived from DTI | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Measurement and instruments are the same as FA. MD describes the overall diffusion and motion of water molecules, with higher MD values reflect more water mobility.
Changes in fractional volume of free water in white matter (FW-WM) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  FW-WM maps were constructed from preprocessed diffusion-weighted images using a regularized bi-tensor model and the open-source software package Diffusion Imaging in Python (also known as Dipy) algorithm (https://dipy.org/). Elevated FW -WM suggests the stagnation of fluid drainage caused by glymphatic dysfunction.
Changes in diffusion tensor image analysis along the perivascular space (DTI-ALPS) index | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The ALPS index was analyzed on DTI images using a method developed and validated by Taoka et al. ALPS index = (mean (Dxxproj, Dxxassoc)) ∕ (mean (Dyyproj, Dzzassoc)). The ALPS indices in the bilateral hemispheres were calculated, respectively, and the mean was used in further analyses. The DTI-ALPS index is calculated from the diffusivity along the deep medullary vein at the level of the lateral ventricle body, as a measure of perivascular clearance activity in the human brain. It is validated as a non-invasive proxy for glymphatic functioning, with higher value indicating better function.
Changes in perivascular space volume fraction in white matter (PVSVF-WM) | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  PVSs were mapped from T2W images using an automated and highly reliable quantification method, following the pipeline of previous studies. The PVS volume fraction (PVSVF) = PVS volume/intracranial volume. The PVSVF-WM is a quantitative metric that reflects the distribution and dilatation of perivascular spaces within cerebral white matter. An elevated volume fraction may suggest impaired clearance function of brain interstitial fluid.
Changes in functional MRI-derived odor-induced brain activation | from baseline to the 48 weeks of treatment.
  Task-evoked activation was assessed using FSL FEAT (version 6.0.7), which use general linear modelling to estimate scent effects on brain activation. Bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, and hippocampus in Automated Anatomical Labeling templates and Brodmann areas 28 and 34 (entorhinal cortices) were extracted and merged as olfactory regions of interest (ROIs) (total cluster size 5,029 voxels) for further analyses.
Changes in plasma amyloid beta (Aβ)42/Aβ40 concentration | from baseline to the 48 weeks of treatment.
  Plasma Aβ40 and Aβ42 concentration were measured using the Neurology 4-plex E assay kit from Quanterix.
Changes in plasma phosphorylated tau (p-tau)181 concentration | from baseline to the 48 weeks of treatment.
  Plasma p-tau 181 concentration was measured using the p-Tau181 Advantage PLUS kit from Quanterix.
Changes in plasma p-tau 217 concentration | from baseline to the 48 weeks of treatment.
  Plasma p-tau 217 concentration was measured using the ALZpath p-Tau217 Advantage PLUS kit from Quanterix.
Changes in plasma neurofilament light chain (NfL) concentration | from baseline to the 48 weeks of treatment.
  Plasma NfL concentration was measured using the Neurology 4-plex E assay kit from Quanterix.
Changes in plasma glial fibrillary acidic protein (GFAP) concentration | from baseline to the 48 weeks of treatment.
  Plasma GFAP concentration was measured using the Neurology 4-plex E assay kit from Quanterix.
Changes in resting-state functional MRI-derived brain network connectivity | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The whole-brain network functional connectivity analysis was carried out using the CONN Toolbox (v.22.v2407). The Schaefer-Yeo 7-network functional atlas was used to parcellate the cortex into 400 volumetric functional parcels, and the Melbourne Subcortical Atlas was used to parcellate the subcortex into 54 functional nuclei, yielding a total of 454 regions. For each participant, the pre-processed resting-state fMRI time series was spatially averaged across all voxels composing each region, yielding an averaged time series for each region. The Pearson correlation coefficient was computed between all pairs of regions from the combined cortical and subcortical atlases to provide a measure of functional connectivity, yielding a 454*454 symmetric connectivity matrix for each individual.
Changes in olfactory threshold scores | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Olfactory Function Assessment by Computerized Testing (OLFACT®, Osmic Enterprises, Inc.) was administered to assess olfactory threshold, identification, and memory. The olfactory threshold test (score range, 1-14) was a forced-choice paradigm based on serial dilutions of N-butanol solutions. Higher scores indicate better olfactory function.
Changes in olfactory identification scores | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Olfactory Function Assessment by Computerized Testing (OLFACT®, Osmic Enterprises, Inc.) was administered to assess olfactory threshold, identification, and memory. The olfactory identification (score 0-30) and memory (score 0-20) subtests consisted of two sequential phases separated by a 10-min interval. During task A, participants performed forced-choice identification of 10 distinct odors. In task B, they were presented with 20 odors (10 from task A and 10 novel distractors) and required to complete two tasks per odor: identify the odor, then classify it as 'old' or 'new' (relative to task A). Higher scores indicate better olfactory function.
Changes in olfactory memory scores | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Olfactory Function Assessment by Computerized Testing (OLFACT®, Osmic Enterprises, Inc.) was administered to assess olfactory threshold, identification, and memory. The olfactory identification (score 0-30) and memory (score 0-20) subtests consisted of two sequential phases separated by a 10-min interval. During task A, participants performed forced-choice identification of 10 distinct odors. In task B, they were presented with 20 odors (10 from task A and 10 novel distractors) and required to complete two tasks per odor: identify the odor, then classify it as 'old' or 'new' (relative to task A). Higher scores indicate better olfactory function.
Changes in olfactory assessment total scores | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  The sum of the olfactory threshold, identification, and memory scores was referred to as the olfactory assessment total scores, which ranged from 0 to 64 points. Higher scores indicate better olfactory function.
Change in glycated haemoglobin (HbA1c) levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Glycated haemoglobin A1c (HbA1c).
Change in fasting plasma glucose levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting plasma glucose.
Change in 2-hour postprandial plasma glucose levels | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  2-hour postprandial plasma glucose.
Change in fasting insulin | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting insulin.
Change in fasting C-peptide levels | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting C-peptide levels.
Change in 2-hour postprandial insulin | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  2-hour postprandial insulin.
Change in 2-hour postprandial C-peptide levels | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  2-hour postprandial C-peptide levels.
Change in pancreatic islet function (HOMA2-β) | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Pancreatic islet function (HOMA2-β) was estimated from fasting C-peptide via HOMA2 Calculator (v2.2.3, http://www.dtu.ox.ac.uk/homacalculator/) .
Change in insulin sensitivity (HOMA2-S) | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Insulin sensitivity (HOMA2-S) was estimated from fasting C-peptide via HOMA2 Calculator (v2.2.3, http://www.dtu.ox.ac.uk/homacalculator/) .
Change in insulin resistance indexes (HOMA2-IR) | from baseline to weeks 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Insulin resistance indexes (HOMA2-IR) was estimated from fasting C-peptide via HOMA2 Calculator (v2.2.3, http://www.dtu.ox.ac.uk/homacalculator/) .
Change in fasting serum triglyceride levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting serum triglyceride levels
Change in fasting serum total cholesterol levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting serum total cholesterol levels
Change in fasting serum high-density lipoprotein-cholesterol levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting serum high-density lipoprotein-cholesterol levels
Change in fasting serum low-density lipoprotein-cholesterol levels | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Fasting serum low-density lipoprotein-cholesterol levels
Change in visceral fat area | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Visceral fat area was measured by Inbody 720 analyser.
Change in percent body fat | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Percent body fat was measured by Inbody 720 analyser.
Change in liver stiffness | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Liver stiffness measurement was quantified by FibroTouch® system
Change in liver fat controlled attenuation parameter | from baseline to weeks 24, 48, and 76 of treatment (the core study spans from baseline to 24, and 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Liver fat controlled attenuation parameter was quantified by FibroTouch® system
Change in blood pressure | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Systolic and diastolic blood pressure
Change in body weight | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Body weight
Change in body mass index | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Body mass index
Change in waist circumference | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Waist circumference
Change in hip circumference | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Hip circumference
Change in waist to hip ratio | from baseline to week 48. (Measurements will be performed every 8 weeks until week 76, with data collected after week 48 will be analyzed and reported after the extension phase).
  Waist circumference to hip circumference ratio
Changes in Barthel index | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Basic activities of daily living (BADL) ability measured by the Barthel index. The Barthel Index (Chinese version) measures dependence in 10 basic personal activities of daily living such as showering, feeding, and walking. Ten items are rated, for a maximum score of 100 representing total independence. A "good" score is ≥ 60 points, which indicates that the patient is capable of basic self-care. Moderate dysfunction is defined as a score between 40 and 60, indicating that the patient needs help in daily life. Severe dysfunction is defined as a score between 20 and 40, indicating that the patient is significantly dependent on help in daily living. A score below 20 indicates a total disability in which the patient depends on help for all aspects of daily living. The measure is completed based on input from the direct care worker providing care to the participants on the day testing.
Changes in FAQ score | from baseline to week 48, and 76 of treatment (the core study spans from baseline to 48 weeks, and the week 76 assessment will be analyzed and reported after the extension phase).
  Instrumental activities of daily living (IADL) ability measured by FAQ scores. The Functional Activities Questionnaire (FAQ, Chinese version) is a standardized assessment of instrumental activities of daily living such as preparing balanced meals and managing personal finances. Sum scores range from 0 to 30, with higher scores indicating worse function. Functional dependence is considered with scores ≥5 points.
Mild cognitive impairment (MCI) remission rate at week76 | from baseline to week 76 of treatment (the week 76 assessment will be analyzed and reported after the extension phase).
  MCI mitigation is defined by three criteria: an education-adjusted score of the Montreal Cognitive Assessment (MoCA) ≥26, no cognitive deficits in any explored cognitive subdomain, including processing speed, executive function, immediate memory, visuospatial construction ability, language, attention and delayed memory, evaluated by Trail-Making Test, Stroop Color-Word Test and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), respectively, and preservation of ability to perform instrumental activity of daily living (IADL) with a Functional Activities Questionnaire (FAQ) score <5.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, MD, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (5):
- China (5):
  - Department of Endocrinology, Changzhou No.2 People's Hospital, the Affiliated Hospital of Nanjing Medical University, Changzhou, Jiangsu
  - Department of Endocrinology, Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Department of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Department of Endocrinology, the Affiliated Jiangning Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Department of Endocrinology, The Affiliated Wuxi People's Hospital of Nanjing Medical University, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Data Availability:
  De-identified participant data may be shared with qualified researchers upon request, subject to review and approval.
  Access Conditions:
  Data requests require a valid research proposal and signed data use agreement. Approval is contingent on compliance with applicable laws and ethical guidelines.
  Timing:
  Data will become available after study completion and primary publication.
  Restrictions:
  Certain data types may be excluded due to privacy or regulatory requirements.
  Contact:
  Requests should be submitted to the study sponsor for consideration.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after study completion and primary publication for 3 years.
Access Criteria: Data requests require a valid research proposal and signed data use agreement. Approval is contingent on compliance with applicable laws and ethical guidelines.

REFERENCES:
- [Result] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697
- [Result] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Lu J, Bi Y, Zhu D. Altered Odor-Induced Brain Activity as an Early Manifestation of Cognitive Decline in Patients With Type 2 Diabetes. Diabetes. 2018 May;67(5):994-1006. doi: 10.2337/db17-1274. Epub 2018 Mar 2. PMID 29500313
- [Result] Cheng H, Zhang Z, Zhang B, Zhang W, Wang J, Ni W, Miao Y, Liu J, Bi Y. Enhancement of Impaired Olfactory Neural Activation and Cognitive Capacity by Liraglutide, but Not Dapagliflozin or Acarbose, in Patients With Type 2 Diabetes: A 16-Week Randomized Parallel Comparative Study. Diabetes Care. 2022 May 1;45(5):1201-1210. doi: 10.2337/dc21-2064. PMID 35263425
- [Derived] Yu C, Yang H, Zhang B, Chen S, Yang S, Li F, Zhu W, Zhai B, Wu T, Zhao S, Zhang W, Tong X, Duan Y, Zhang L, Chao Y, Wu J, Zhu X, Wang K, Ye X, Zhang X, Xu X, Cheng H, Liu J, Zhang J, Wang Y, Zhang Z, Yan W, Bi Y. Evaluating the effects of liraglutide, empagliflozin and linagliptin on mild cognitive impairment remission in patients with type 2 diabetes (LIGHT-MCI): study protocol for a multicentre, randomised controlled trial with an extension phase. BMJ Open. 2025 Aug 21;15(8):e095382. doi: 10.1136/bmjopen-2024-095382. PMID 40840993
- Available data/document: Statistical Analysis Plan: 10.6084/m9.figshare.30994510 — https://figshare.com